CLINICAL TRIAL: NCT03628170
Title: Evaluation of the Soft Tissue Profile Following Socket Preservation With Platelet Rich Fibrin Versus Free Gingival Graft: A Randomized Controlled Study
Brief Title: Soft Tissue Profile Following Socket Preservation With Platelet Rich Fibrin Versus Free Gingival Graft
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Haya Hesham, Principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: version 3
Record Dates: First submitted 2018-05-04; First posted 2018-08-14 (Actual); Last update posted 2018-08-14 (Actual); Status verified 2018-05

CONDITIONS: Soft Tissue Mass

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRF (Platelet -rich fibrin) group (Experimental): Extraction of the tooth followed by Platelet rich fibrin placed in the socket covered bu platelet rich fibrin membrane for socket preservation.
  Interventions: Other: platelet rich fibrin
- Free gingival graft group (Active Comparator): Extraction of the tooth followed by using free gingival graft to cover the socket for socket preservation.
  Interventions: Other: Free gingival graft

INTERVENTIONS:
Other: platelet rich fibrin — platelet rich fibrin will be prepared from patient's venous blood and inserted in the centrifuge at 2000 r.p.m. for 12 minutes Then, the Platelet rich fibrin plug will be placed in the socket after extraction for socket preservation covered by platelet rich fibrin membrane.
  Arms: PRF (Platelet -rich fibrin) group
Other: Free gingival graft — Free gingival graft will be taken from the palate to cover the socket after extraction of the tooth for socket preservation.
  Arms: Free gingival graft group

SUMMARY:
Comparing socket preservation with Platelet -Rich Fibrin versus Free gingival graft.

DETAILED DESCRIPTION:
Extraction of the non restorable tooth, then socket preservation is applied in experimental group using platelet rich fibrin, while in comparative group free gingival graft is applied with socket preservation.

ELIGIBILITY:
Inclusion Criteria:

* Age range 25-50 years.
* Non- restorable teeth indicated for extraction.
* Good oral hygiene.
* Intact facial and lingual plates of bone, without infection or pathosis.
* Adequate apiacl bone for primaru stability

Exclusion Criteria:

* Presence of uncontrolled Systemic disease eg: diabetes, bone disease or the use of medicines that interfere with bone metabolism, history of head and neck radiotherapy.
* Presence of periodontal and/or periapical infection.
* Smokers.
* Non-compliant patients.
* Pregnancy or lactation in females.
* History of head and neck radiotherapy.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2018-06-07 (Actual); Primary Completion 2019-01 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Soft tissue profile change | 6 months
  Optical scanning by optical scanner at baseline to the preoperative cast of the related area, then optical scanning to postoperative cast of the surgical area after 6 months. Then, superimposition between the two scans of the casts will be performed to measure the difference or change in the amount of soft tissue profile measured in millimeters between baseline and at 6 months

SECONDARY OUTCOMES:
Crestal bone level change | 6 months
  measured by Cone beam computed tomography (CBCT) taking the neighboring teeth as reference points, with superimposition between readings at baseline and at 6 months.
  Superimposition will identify the difference or change in crestal bone level measured in millimeters between baseline and at 6 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Oral and dental medicine, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
After reaching for the primary and secondary outcomes, international publication will be performed